CLINICAL TRIAL: NCT04092192
Title: Prospective Comparison of Rigid Forceps Versus Endovascular Snare for Routine IVC Filter Retrieval
Brief Title: Forceps vs. Snare IVC Filter Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB 18-1502
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: DVT
Keywords: IVC filter, filter removal, filter retrieval

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Forceps (Active Comparator): Subjects randomized to this cohort will have their IVC filter removed using a rigid forceps device that will be used to engage the filter apex directly and allow for the filter to be capture/removed.
  Interventions: Device: IVC filter removal
- Snare (Active Comparator): Subjects randomized to this cohort will have their IVC filter removed using an endovascular snare (like a lasso) device that is designed to catch the hook of the filter and allow it to be captured.
  Interventions: Device: IVC filter removal

INTERVENTIONS:
Device: IVC filter removal — In the clinic, it will be explained to patient that they are asked to participate in a study that would randomize them to one of two established techniques for IVC filter removal. It will be explained these are both techniques that are used by interventional radiologists normally used for IVC filter retrieval.
  One technique would be the utilization of an endovascular snare (like a lasso) device that is designed to catch the hook of the filter and allow it to be captured.
  The other technique described will be the usage of a rigid forceps device that will be used to engage the filter apex directly and allow for the filter to be capture/removed.

SUMMARY:
IVC filters are mechanical filters placed in a patient's body to trap blood clots in the legs migrating to the lungs. When no longer indicated, interventional radiologists are consulted for IVC filter removal. Currently, many methods for extracting IVC filters exist. Two of the most common methods involve using an endovascular snare device or rigid forceps. We intend to prospectively compare these two methods in an attempt to see if one offers an advantage to the other. This will be compared by evaluating success rates and procedure time.

DETAILED DESCRIPTION:
Currently the optimal method for IVC filter retrieval with respect to success rate and fluoroscopic time (i.e. radiation exposure) is poorly understood. Both snare and forcep techniques have independently evaluated in literature but have never been compared directly. The proposed study would prospectively assess whether one of these established technique offers an advantage with respect to either of these variables.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant females
* Adult patients (age 18 years and older)
* Referred to Interventional Radiology for IVC filter removal
* IVC filter implanted less than 6 months with the procedure being performed at UCMC by current IR staff.
* Cook Celect filter or Argon Medical Option Elite

Exclusion Criteria:

* Patients with outside hospital filter placement
* Filters other than Cook Celect or Argon Medical Option Elite
* Implantation period >6 months
* Evidence of coagulopathy (INR <1.8, platelet count >50k)
* Clotting disorder
* Central venous occlusion
* Prior filter placement/removal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-26 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Removal success rate | Procedure date
  Data will be analyzed by a biostatistician to determine statistical differences between cohorts with respect to outcome measures.
Flouroscopy time | Procedure start to finish
  Venography will be performed using a flush catheter and contrast material to evaluate for tip embedding. After filter retrieval, repeat venography will be performed to evaluate for thrombosis, caval spasm, caval perforation, fractured fragments, and other potential complications.
Costs | Date of procedure up through 6 months following IVC filter removal
  Costs associated with filter removal encounter
Procedure related complications | Date of procedure through 6 months following IVC filter removal
  After hemostasis is achieved, patients will be monitored for 2-4 hours in the interventional radiology recovery area.
  One month after filter retrieval, patients will be seen in clinic for follow-up. During this visit, a physicial assessment will done, including adverse events and review of medications.
  Six months after filter retrieval, patient will be contacted by telephone for follow-up. Adverse event and medication review will be performed during this call.

CONTACTS AND LOCATIONS:
Overall Officials: Osmanuddin Ahmed, MD, Principal Investigator — UChicago Medicine
Locations (1):
- UChicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared